CLINICAL TRIAL: NCT05351138
Title: Comparison the Efficiency of Transcutaneous Electrical Nerve Stimulation and Manual Therapy in Children With Cerebral Palsy With Lower Urinary System Dysfunction
Brief Title: Comparison of Transcutaneous Electrical Nerve Stimulation and Manual Therapy in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Collaborators: Tugtepe Pediatric Urology Clinic (Other)
Responsible Party: Principal Investigator, Pelin Pişirici, Assistant Professor, PT, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BBD-TUGTEPE-130422
Record Dates: First submitted 2022-04-13; First posted 2022-04-28 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Bladder Dysfunction; Bowel Dysfunction; Cerebral Palsy; Neurogenic Bladder; Neurogenic Bowel
Keywords: Neuromodulation therapy; Urinary incontinence; Constipation; Voiding disorder; Abdominal massage
MeSH Terms: conditions — Intestinal Diseases; Cerebral Palsy; Urinary Bladder, Neurogenic; Neurogenic Bowel; Urinary Incontinence; Constipation | interventions — Transcutaneous Electric Nerve Stimulation; Massage

STUDY DESIGN:
Intervention Model Description: Children between the ages of 5-18, diagnosed with CP with LUTD who met the inclusion criteria will be included in the study. Sample size of the study is calculated as 54. All evaluations of the participants will be done by the specialist physiotherapist who made the evaluations would not know which treatment method was applied to the participants and would be a blind evaluator.
Who Masked: Outcomes Assessor
Masking Description: The children to be included in the study will be randomized into two groups as the TENS group (TG) and the massage group (MG) after the first day evaluations are completed. Randomization will be done with the www.randomizer.com site. The groups of children determined according to the order of participation will be placed in opaque envelopes and the envelopes will be closed. On the second day, the physiotherapist, who will apply the treatments, will do the application according to the group that comes out of the envelope.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS Group (Experimental): Transcutaneus electric nerve stimulation intervention will be done for a total of 12 weeks, 2 sessions of 20 minutes per week.
  Interventions: Device: TENS
- Masaj Group (Experimental): Massage intervention will be done in the form of massage practise to the abdominal region, 2 sessions of 20 minutes per week.
  Interventions: Other: Massage

INTERVENTIONS:
Device: TENS — In the study, CE certified tens device with Biolito brand, which is used specifically for incontinence treatment, will be used. The electrodes used during the intervention will be placed to the parasacral region (S2-S4). While the current is given, the power of the device will be gradually increased in 1 mA intervals. The lower value of the stimulation will be 10 mA and the upper value will be 25 mA, and the treatment will be continued with any value that the child can tolerate in this range.
  Arms: TENS Group
Other: Massage — The massage will be applied to the abdominal area between the subcostal lower border and the anterior superior of the spina iliaca. Massage techniques are as follows: Abdominal patting, colon patting, colon kneading, colon patting again, abdominal patting again. It will be advanced with deep abdominal strokes, then the starting point will be returned with transverse superficial strokes for the transversus abdominis muscle and oblique superficial strokes for the rectus abdominis muscle, and these strokes will be repeated 3 times each, a total of 6 times. Afterwards, 3 times column brushing, 3 times column kneading and 3 times column plastering will be done, respectively. At the end, a total of 6 abdominal strokes will be performed for both the transversus abdominis and oblique abdominal muscles as in the beginning.
  Arms: Masaj Group

SUMMARY:
There are many studies in the literature on healthy children with lower urinary tract dysfunction (LUTD), but there are limited number of studies in children with cerebral palsy (CP) with LUTD.

This study aim to contribute to the literature by examining the effectiveness of transcutaneous electrical nerve stimulation (TENS) and abdominal massage in the treatment of children with CP with LUTD and comparing the superiority of the two treatment methods to each other.

DETAILED DESCRIPTION:
CP represents a group of chronic, non-progressive motor disorders characterized by impaired voluntary movement resulting from prenatal developmental abnormalities or perinatal or postnatal central nervous system damage.

The location and extent of neurological damage are important in determining motor and mental disabilities and the severity of the disease. Children with CP can also be affected by other medical disorders such as seizures, mental retardation, hearing, vision and communication problems. The prevalence of CP is approximately 2-3 per 1000 live births. Dysfunctional bowel and urinary dysfunction problems can often accompany CP due to motor, mental, cognitive, sensory and other neurological disorders. Severe motor disorders and/or additional cognitive deficits lead to the development of neurogenic lower urinary tract symptoms. Accoring the data obtained during the outpatient clinic visits, it was determined that most of the children with CP had LUTD complaints such as incontinence, sense of urgency, difficulty urinating, urinary retention and urinary tract infections. These urological problems affect approximately one-third of children with CP, and the prevalence of dysfunctional voiding symptoms such as pollakisuria, incontinence or urinary tract infections is estimated to be more than 30% in the population.

TENS therapy is classified as a neuromodulation therapy. In the last few years, it has been shown in the literature TENS gives positive results in the treatment of urinary symptoms.

Abdominal massage, which is one of the manual therapy techniques; the anterior abdominal wall reduces abdominal muscle tension, increases local circulation, facilitates digestion and stimulates gastric acid secretion, stimulates colonic movements by providing peristaltic stimulation. It is a classical massage method that includes clockwise manual movements over the area where the colon is located. In abdominal massage, by manually applying pressure from the anterior abdominal wall, the digestive organs are compressed between the fingers and the posterior abdominal wall and peristaltic stimulation is created. Hence, stool is pushed from the colon into the rectum. In addition, abdominal massage reduces the severity of constipation symptoms by reducing abdominal bloating and treating trigger points in the abdominal muscles.

This study aim to contribute to the literature by examining the effectiveness of TENS and abdominal massage in the treatment of children with CP with LUTD and comparing the superiority of the two treatment methods to each other.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 5-18
* Diagnosed with Cerebral Palsy
* Having one of the Gross Motor Function Classification System I, II, III and IV grades
* Having a complaint of urinary incontinence

Exclusion Criteria:

* Being younger than 5 years old
* Being level V according to Gross Motor Function Classification System
* Having uncontrolled epileptic seizures
* Anatomical changes in the urinary system
* Having cognitive disability

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Voiding Disorders Symptom Scoring | Change from Baseline at 12th week
  Voiding Disorders Symptom Scoring was developed in 2005 and includes 13 questions about symptoms and 1 question about quality of life .
  The scale is for parents and scoring is done according to the answers from the parents. The total score is between 0-35 points. As the score obtained from the scale increases, the severity of the patient's symptoms also increases.

SECONDARY OUTCOMES:
Bladder Diary | Change from Baseline at 12th week
  The bladder diary is a simple and non-invasive method of assessing people with lower urinary tract symptoms. The International Children's Continence Society has proposed a chart to assess lower urinary tract dysfunction, showing 48-hour daytime voiding frequency, voiding volume, voiding duration, presence of urgency, type and amount of fluid intake, and degree of urinary incontinence.
Pediatric Incontinence Quality of Life Scale | Change from Baseline at 12th week
  Pediatric Incontinence Quality of Life Scale is the first continence quality of life scale developed in the pediatric population. It is a continence-specific quality of life scale developed for children and adolescents in 2006. The Turkish validity and reliability study was performed in 2011.
  In the initial development stages of the PINQ scale, it was developed as 28 questions including 7 dimensions that evaluate children's social relations with their peers, self-esteem, family and home relations, body image, independence, mental health and treatment. In the following studies, these dimensions were grouped into two as Extrinsic (extrinsic) and Intrinsic (intrinsic), and finally the number of questions was arranged as 20. Each question is given a score of 0 (no), 1 (almost never), 2 (sometimes), 3 (often), 4 (always), and a total score (0-80) is calculated. An increase in the total score indicates that the patient's quality of life worsens .
Rome IV Criteria | Change from Baseline at 12th week
  Rome IV criteria allow to detect the presence of constipation in toilet trained or untrained children. Abdominal pain that recurs at least once a week in the last 3 months; If defecation is associated with at least two of the symptoms of a change in the frequency of pooping and a change in the form of poop, constipation is present according to the Rome 4 criteria.
Bristol Stool Scale | Change from Baseline at 12th week
  The Bristol Stool Scale (BSS) was developed by Lewis and Heaton at the University of Bristol in 1990 and classifies human faeces into 7 groups. The shape of the stool changes according to the time it stays in the colon. The BSS is a fast and reliable indicator of transit time. There are 7 different poop forms on the Bristol stool scale. Types 3 and 4 correspond to the normal poop form. Types 1 and 2 show that the person has symptoms of constipation. Tip 5,6,7 corresponds to (in order) lack of fiber, mild diarrhea and severe diarrhea.

CONTACTS AND LOCATIONS:
Overall Officials: Betül Ünal, PT, Principal Investigator — Bahçeşehir University, Graduate Education Institute, Physical Therapy and Rehabilitation; Pelin Pişirici, PT, PHD, Study Director — Bahçeşehir University, Health Sciences Faculty, Physiotherapy and Rehabilitation Department; Halil Tuğtepe, MD, Prof., Study Chair — Private Tuğtepe Pediatric Urology and Surgery Clinic; Aygül Köseoğlu, PT, Msc, Study Chair — Private Tuğtepe Pediatric Urology and Surgery Clinic
Locations (1):
- Pelin Pişirici, Istanbul, Besiktas/Istanbul, Turkey (Türkiye)